CLINICAL TRIAL: NCT00003569
Title: Phase I Trial of Escalating Doses of BNP7787 in Patients With Solid Tumors Undergoing Treatment With Cisplatin and Taxol
Brief Title: Dimesna in Treating Patients With Solid Tumors Who Are Undergoing Treatment With Cisplatin and Paclitaxel
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: DS 97-39; RPCI-DS-9739; BIONUM-BNP7787IV101; NCI-G98-1478
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Head and Neck Cancer; Lung Cancer; Neurotoxicity; Ovarian Cancer
Keywords: stage III non-small cell lung cancer; recurrent non-small cell lung cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage IV non-small cell lung cancer; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; neurotoxicity; recurrent salivary gland cancer; stage IV salivary gland cancer; salivary gland squamous cell carcinoma; stage III salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Neurotoxicity Syndromes; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Cisplatin; 2,2'-dithiodiethanesulfonic acid; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: dimesna
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as dimesna may protect normal cells from the side effects of chemotherapy.

PURPOSE: This phase I trial is studying the side effects and best dose of dimesna in treating patients with solid tumors who are receiving cisplatin and paclitaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of dimesna administered prior to cisplatin and paclitaxel in patients with solid tumors.
* Determine the dose related qualitative and quantitative side effects of dimesna administered on this schedule in these patients.
* Determine the minimum safe volume of intravenous hydration after the determination of the MTD of dimesna in these patients.
* Investigate the possible protective side effects of dimesna in reducing or preventing the development of cisplatin induced nephrotoxicity and observe possible protective effects against cisplatin or paclitaxel related neurotoxicity and myelosuppression in these patients.
* Investigate the pharmacokinetic behavior of dimesna in the plasma and urine on this schedule of administration in this patient population.

OUTLINE: This is a dose-escalation, two-stage, multicenter study.

During stage I, patients receive a single dose of dimesna IV over 15 minutes 7 days prior to chemotherapy. Patients then receive paclitaxel IV over 3 hours followed by dimesna IV over 15-30 minutes followed immediately by cisplatin IV over 1 hour on day 1 every 3 weeks. Patients continue courses of paclitaxel, dimesna, and cisplatin every 3 weeks in the absence of disease progression or unacceptable toxicity for up to 6 courses.

In stage I, cohorts of 3-6 patients each receive escalating doses of dimesna until the maximum tolerated dose (MTD) is reached. The MTD is defined as the highest dose at which no more than 1 of 6 patients experiences dose limiting toxicity (DLT). The MTD of dimesna is then used in stage II of the study, in which the volume of pre and post cisplatin intravenous saline hydration is reduced in cohorts of 3-6 patients each. The MTD intensity of cisplatin is defined as the least saline hydration volume at which no more than 1 of 6 patients experience DLT.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer, ovarian carcinoma, squamous cell carcinoma of the head and neck, tumor types for which no standard treatment exists, or tumor types that have failed standard therapy
* Paclitaxel and cisplatin combination therapy must be an appropriate option in treating disease
* No potentially curable type of cancer (e.g., newly diagnosed testicular cancer)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 6 weeks

Hematopoietic:

* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT and SGPT normal

Renal:

* Creatinine normal
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No evidence of congestive heart failure
* No uncontrolled moderate to severe hypertension
* Includes patients with persistent elevated systolic blood pressures of greater than 170 mm Hg and diastolic blood pressures of greater than 100 mm Hg for more than 1 month while under medical treatment

Other:

* No active infection
* No perceived or actual clinical risk of cisplatin induced toxicity that exceeds the clinical benefit of using cisplatin therapy
* No known history of severe hypersensitivity to polyoxyl 35 castor oil vehicle
* No severe medical problems unrelated to malignancy that would interfere with compliance in this study
* Not pregnant
* Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent colony stimulating factors except for febrile neutropenia
* No concurrent aminoglycoside therapy except for febrile neutropenia or other life threatening infections
* No concurrent immunotherapy

Chemotherapy:

* At least 6 weeks since prior nitrosoureas or mitomycin
* At least 3 weeks since other prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to measurable disease

Surgery:

* At least 2 weeks since prior major surgery

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 1998-03; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Creaven, MBBS, PhD, Study Chair — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York